CLINICAL TRIAL: NCT05054322
Title: A Multicenter, Open-label, Randomized Controlled Trial to Evaluate the Efficacy of Fluticasone Propionate MDI Added to Standard Care at Early Stage of COVID-19 in Reducing the Incidence of Adverse Outcomes in Symptomatic Patients Either From 18 to 49 Year Old With Risk Factors or Older Than 50 Year Old
Brief Title: FLuticasone in cOvid Treatment (FLOT)
Acronym: FLOT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Vu Tran Thien Quan, Lecturer, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 466/HDDD-DYHD
Record Dates: First submitted 2021-09-20; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: COVID19; Fluticasone Propionate; inhaled corticosteroid; ICS
MeSH Terms: conditions — COVID-19 | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants will be monitored via video call twice a day without any specific drugs.
- Fluticasone propionate with spacer (Experimental): Fluticasone propionate 125 mcg with spacer, 4 puffs, twice a day, added to standard care
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate — Fluticasone propionate added to usual care, total dose 1000 mcg per day for 14 days
  Other Names: Flixotide 125 mcg Evohaler
  Arms: Fluticasone propionate with spacer

SUMMARY:
A multicenter, open-label, randomized controlled trial to evaluate the efficacy of fluticasone propionate (metered dose inhaler - MDI) added to standard care at early stage of COVID-19 in reducing the incidence of adverse outcomes (any of those following: oxygen therapy, systemic corticosteroids, hospitalization, mechanical ventilation, and mortality) in symptomatic patients either from 18 to 49 years of age with risk factors or older than 50 years.

DETAILED DESCRIPTION:
This study has 2 arms: the standard care group followed the COVID-19 guidelines of the Ministry of Health of Vietnam and the interventional group: Fluticasone propionate MDI with spacer, twice a day for 14 days.

The study participants will be monitored via video call from day 1 to day 14, day 21, and day 28 after randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Signing consent to participate in the study
2. Having COVID related-symptoms within 5 days prior to randomization
3. Confirmed diagnosis of COVID-19 by rapid antigen test or polymerase chain reaction (PCR) test within 5 days prior to randomization
4. Over 50 years old OR 18-49 years old and have one or more of risk factors for severe COVID-19

Exclusion Criteria:

1. Pregnant or breastfeeding woman
2. Allergy and/or contraindications to inhaled Fluticasone
3. Current or previous administration of inhaled corticosteroids within the 15 days prior to randomization
4. Current or previous administration of high dose systemic corticosteroids (higher than 3.75 mg dexamethasone/day or equivalent doses of other corticosteroids) and/or anticoagulants etc.. more than or equal to 2 days within 15 days prior randomization, or taking any other antiviral drugs (such as remdesivir, favipiravir, etc..)
5. Indication for start of systemic corticosteroids or oxygen therapy or hospitalization dut to COVID-19 within next 24 hours
6. Already participated in other interventional COVID studies
7. Any conditions for which the investigator believes that the patient should not participate for the benefit of the patient or that would prevent, limit, or distort the evaluation of the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-09-22 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse outcomes | Day 28 after randomization
  To evaluate the efficacy of fluticasone propionate MDI added to standard care at an early stage COVID-19 in reducing the incidence of adverse outcomes (oxygen therapy, systemic corticosteroids, hospitalization, mechanical ventilation, and mortality) in symptomatic patients either from 18 to 49-year-old with risk factors or older than 50-year-old.

SECONDARY OUTCOMES:
Duration of isolation based on WHO's criteria | Day 28 after randomization
  To evaluate the efficacy of fluticasone propionate MDI added to standard care at early stage COVID-19 in reducing duration of isolation bases on WHO's criteria in symptomatic patients either from 18 to 49-year-old with risk factors or older than 50-year-old
The incidence of patients with oxygen saturation by pulse oximetry (SpO2) <94% | Day 28 after randomization
  To evaluate the efficacy of fluticasone propionate MDI added to standard care at an early stage COVID-19 in reducing the incidence of patients with SpO2<94% in those either from 18 to 49-year-old with risk factors or older than 50-year-old
Self-reported recovery rate | Day 28 after randomization
  To evaluate the efficacy of fluticasone propionate MDI added to standard care at an early stage COVID-19 in reducing self-reported recovery rate of symptomatic patients either from 18 to 49-year-old with risk factors or older than 50-year-old

CONTACTS AND LOCATIONS:
Overall Officials: Thi Tuyet Lan Le, Ph.D., M.D., Principal Investigator — tuyetlanyds@gmail.com
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From Oct 2021 to September 2022.
Access Criteria: Researchers who proposed use of data has been approved by a review committee.